CLINICAL TRIAL: NCT05076994
Title: The PET Project: Patient Education Tool for Home Exercise
Acronym: PET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Steven Macaluso, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 119395
Record Dates: First submitted 2021-08-10; First posted 2021-10-13 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Low Back Pain; Greater Trochanteric Pain Syndrome
Keywords: Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: Two Randomized Groups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education Tool (Experimental)
  Interventions: Other: Exercise therapy
- Standard Care (Active Comparator)
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Exercise therapy — A series of home exercise videos to improve patient adherence to exercise prescription
  Arms: Patient Education Tool
Other: Standard Care — An exercise prescription and verbal instructions in clinic
  Arms: Standard Care

SUMMARY:
Patients presenting to an musculoskeletal (MSK) outpatient clinic who fit the study inclusion criteria (low back pain, outer hip pain) will be randomized to receive an exercise prescription with patient education alone, or in clinic patient education and access to the Patient Education Tool (Series of videos). Weekly surveys will be done via email to assess patient adherence: the main outcome. Two follow-up in-clinic visits at weeks 6 and 12 will assess pain, function and exercise self-efficacy: the secondary outcomes. Comparisons will be made between the group of the patients who received the videos and those who did not.

DETAILED DESCRIPTION:
Musculoskeletal conditions are a very common, if not the most common, reason to visit the family doctor, comprising an estimated one-in-six to over half6 of all primary care visits. Under this umbrella of musculoskeletal conditions fall many different aliments: this paper will investigate chronic nonspecific low back pain and greater trochanter pain syndrome.

Boasting titles for greatest number of disability-years caused by a disease and most common non-communicable disease, one would hope that researchers and clinicians would thoroughly understand what causes this pervasive morbidity. Unfortunately, when it comes to chronic nonspecific low back pain (CNLBP), no clear pathoanatomic cause is attributed to the symptoms.

Low back pain is localized below the costal margin and above the inferior gluteal folds and is deemed chronic when it lasts for more than 12-weeks. Although most cases of low back pain seem to resolve prior to the 12-week mark, chronic low back pain is responsible for the vast majority of workers' compensation costs. In 90% of cases of chronic low back pain, clinicians cannot pinpoint the etiology, hence the 'non-specific' modifier.

Greater trochanter pain syndrome (GTPS) boasts a slightly less impressive resume - affecting a mere 10% to 25% of the general population. GTPS presents as lateral hip pain, specifically over the greater trochanter, and is worse when lying or bearing weight on that side.

It too has a plethora of potential aetiologies, and although it can be challenging to elucidate lateral hip pain's true etiology this clinical diagnosis comprises of trochanteric bursitis, gluteus medius and minimus tendinopathies, and external coxa saltans (commonly referred to as "snapping hip").

CNLBP and GTPS seem to coexist in about a third of the time and general treatment recommendations are similar. They range from analgesic medication to load management, though because between CNLBP and GTPS, a wide demographic is affected, treatments should be accessible and applicable to the wider population. Exercise therapies generally to meet these criteria. Exercise has also routinely demonstrated to be efficacious, cost-effective and low risk.

A multitude of different exercise modalities have routinely been shown to reduce chronic pain and improve physical function. Furthermore, specific exercises can be leveraged to treat chronic pain of broad aetiologies. Systematic reviews and meta-analyses alike have shown these to hold true in the realm of chronic non-specific low back pain as well. Commonly communicated is the relative paucity of research on GTPS, however, minimizing pain and performing strengthening and stretching exercises for the region appears to be a mainstay of the current therapy.

It is well known that exercise program adherence is a major issue when it comes to exercise interventions. A minimum level of adherence must be obtained for an exercise intervention to be efficacious. And when that level of adherence is attained in patients with CNLPB, exercise-based programs have shown to decrease pain and improve function. Similar results are show in the little amount of research on exercise therapies for GTPS, and in clinical practice it is assumed to be true.

Adherence is higher when people are highly supervised. So it is unsurprising that patients have higher rates of adherence after seeing their physiotherapist for extra 'booster' sessions. However, additional sessions with healthcare providers is not always feasible, due to high costs, poor accessibility, or unavailable providers, amongst other reasons. With the ever-increasing use of technology, though, patients can have somewhat similar care - such as guidance while doing exercises - through pre-recorded online videos. Some preliminary studies suggest that these online videos are able to increase patient adherence.

While many YouTube exercise rehabilitation videos are of high quality, there are also many that are not. This can leave the patient - even with an abundance of online resources - paradoxically without answers: unsure and unable to know what is relevant. Additionally, patients report better trust towards those who adequately understand their medical conditions, such as their healthcare team.

It would then be conceivable that physician-produced videos that are endorsed by the patient's healthcare team would alleviate this issue. Furthermore, it could circumvent the challenges associated with in-person care as well as alleviate some of the pitfalls of sifting through endless YouTube videos. The aim of this study was to investigate whether a patient education tool - an accompanying set of explanatory videos - will increase patient adherence when compared to prescribing an evidence-based, personalized set of exercises without these videos.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* The ability to perform at least 5 of the 10 total exercises, as cleared by the physiatrist
* The willingness to comply with the study criteria for its 12-week duration
* The written informed consent of the participant
* Sufficient English comprehension to understand the questionnaires
* Sufficient English comprehension to consent to the study
* Chronic lower back pain:

  o A history of lower back pain exceeding 3 months
* Greater trochanter pain syndrome:

  * A history of lateral hip pain exceeding 3 months
  * Pain in at least three of the following tests: palpation of the greater trochanter, FABER test, resisted external de-rotation test, modified resisted external de-rotation test

Exclusion Criteria:

* Pregnancy
* Condition that makes the exercising ill advisable, as determined by the physiatrist
* Chronic lower back pain:

  * Known lumbar disc herniation
  * Acute phase of lumbar disc protrusion
  * Known vertebral fractures
  * Known infectious, inflammatory, or malignant diseases of the vertebrae
  * Known presence of severe spinal deformity
* Greater trochanter pain syndrome:

  * Acute hip pathology such as fracture, dislocation, infection, etc.
  * Known diagnosis moderate to severe hip osteoarthritis causing significant range of motion restriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Pain | 0 weeks (Day of entry to trial)
  Change in Visual Analogue Scale (VAS) ("No Pain" on one end of scale (0 out of 100), and "Worse pain you can imagine" on the opposite end of the scale (100 out of 100)
Pain | 6 weeks
  Change in Visual Analogue Scale (VAS) ("No Pain" on one end of scale (0 out of 100), and "Worse pain you can imagine" on the opposite end of the scale (100 out of 100)
Pain | 12 weeks
  Change in Visual Analogue Scale (VAS) ("No Pain" on one end of scale (0 out of 100), and "Worse pain you can imagine" on the opposite end of the scale (100 out of 100)

SECONDARY OUTCOMES:
Exercise Adherence Rate | Number of exercises performed each 1 day (24 hours). Data collected once weekly for 12 weeks via online automated survey.
  Daily log of adherence to the exercise prescribed is recorded by participants and submitted on a weekly basis.
Self efficacy and confidence of participants | 0 weeks (day of entry to program)
  Use of the Self Efficacy in Exercise (SEE) standard survey to determine patients' level of confidence to complete the assigned exercises despite various barriers.
  Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Self efficacy and confidence of participants | 6 weeks
  Use of the Self Efficacy in Exercise (SEE) standard survey to determine patients' level of confidence to complete the assigned exercises despite various barriers. Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Self efficacy and confidence of participants | 12 weeks
  Use of the Self Efficacy in Exercise (SEE) standard survey to determine patients' level of confidence to complete the assigned exercises despite various barriers. Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.

IPD SHARING:
Plan to Share IPD: Undecided